CLINICAL TRIAL: NCT02477163
Title: An Observational Clinical Study to Determine the Effect of Multi-modal Ayurvedic Treatment in the Patients of Chronic Kidney Disease
Brief Title: Ayurvedic Management of Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J.S. Ayurveda College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSAM/IECHR/13-14/362-2
Record Dates: First submitted 2015-06-11; First posted 2015-06-22 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Nephropathy; Hypertensive Nephropathy
Keywords: Nephropathy; Chronic Renal Failure; Chronic Kidney Disease; Chronic Renal Disease; Ayurveda; Herbal treatment
MeSH Terms: conditions — Diabetic Nephropathies; Hypertensive Nephropathy; Kidney Diseases; Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Pre-post design
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single group (Experimental): Patients of chronic renal failure
  Interventions: Other: Ayurveda treatment

INTERVENTIONS:
Other: Ayurveda treatment — 1. Gokshuradi Guggulu (compound Ayurvedic preparation: Gokshura + Guggulu + Triphala + Trikatu + Musta) - 1 g, 3 times in a day after food with warm water.
  2. Varunadi kvath (ingredients: Varuna tvak + Bilva moola + Apamarga + Chitrak moola + Arani + Shigru + Bruhati + Kirattikta + Karanja + Shatavari) - 40 ml 2 times in a day after food.
  3. Rasayan Churna (powder of Gokshura + Amalaki + Guduchi in equal quantities ) - 3 g, 3 times a day with water.
  4. Bhumyamalaki (Tamalaki Rasayan) tablet - 1 g, 2 times in a day after food with water.
  5. Uricare (of Punarvasu Pharmacy, Petlad road, Nadiad) tablet - 1 g, 3 times in a day after food with warm water.
  6. Niruha Basti (procto-colonic administration of ayurvedic medicine) with Punarnavadi kvath (decoction) - in the morning, before one hour of the lunch.

SUMMARY:
The purpose of this study is to determine the effect of multi-dimentional ayurvedic treatment in the patients of various types of chronic kidney disease.

DETAILED DESCRIPTION:
Ayurvedic treatment includes some complex classical herbal formulations and Niruha basti (procto-colonic administration of ayurvedic medicines mainly contained decoction of punarnavadi compound, rocksalt, sesame oil and mixture of some herbal poweders) will be given to the patients of chronic kedney disease who are not on dialysis. Patients of CKD of various etiology will be grouped accordingly and will get the same treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a confirm diagnosis of chronic kidney disease with GFR level < 60mL/min and persistent (present for > 3 months) indicates substantial reduction in kidney function. Confirmation of diagnosis with ultrasound of KUB, indicating reduction of kidney size and / or cortico-medullary difference.

Exclusion Criteria:

* Female patients having pregnancy, breast feeding or post-delivery period.
* Patients who are on dialysis treatment from more than 6 months period. Patients who are already operated for renal transplantation and then having nephropathy.
* Patients with some serious illness like cardio-vascular diseases, acute mental disorders, serious acute organic diseases, serious chronic co-morbidity, hypo or hyper thyroidism, other kidney, liver or metabolic disorders etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Improvement in the signs and symptoms | 4 weeks
  Following grade score will be used to measure the improvement in all the patients at the initial level and after the treatment.
  Grade score of signs and symptoms
  1. Oedema: No oedema(0); Slight oedema on lower extremties(1); Severe oedema on lower extrimities(2); Anasarca(3)
  2. General weakness: No weakness(0); Mild weakness(1); Moderate weakness(2); Severe weakness(3)
  3. Loss of appetite: Good appetite(0) Mild loss of appetite(1); Moderate loss of appetite(2); Complete loss of appetite(3)
  4. Nausea / Vomiting: Absent(0); Occasional(1); Once or twice a week(2); Daily(3)
  5. Muscle cramps: Absent(0); Occasional(1); Once or twice a week(2); Daily(3)
  6. Breathlessness: Absent(0); On fast walking or climbing stairs(1); Sometimes at rest(2); Generally occurs at rest(3)
  7. Hiccup: Absent(0); Occasional(1); Once or twice a week(2); Daily(3)
  8. Pruritus: Absent(0); Mild(1); Moderate(2); Severe(3)
Changes in the value of laboratory investigations | 4 weeks
  All the related laboratory investigations will be done before and after the treatment. Effect will be assessed with the help of reduction level in serum creatinine(in mg /dl), blood urea(in mg/dl), serum uric acid(in mg/dl) and improvement in hemoglobin(in gm%) and serum electrolytes level(in mmol/l).

CONTACTS AND LOCATIONS:
Overall Officials: Manishkumar V Patel, MD(Ayurveda), Principal Investigator — J S Ayurveda College,College Road, Nadiad
Locations (1):
- P D Patel Ayurveda Hospital, Nadiād, Gujarat, India